CLINICAL TRIAL: NCT03873272
Title: Randomized Controlled Selection Trial of Cryotherapy vs. Compression Therapy for the Prevention of Taxane-induced Peripheral Neuropathy in Breast Cancer Patients
Brief Title: The CONTRoL Trial: Cryotherapy vs. cOmpression Neuropathy TRiaL
Acronym: CONTRoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa K Accordino, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: AAAR9515
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy
Keywords: Neuropathy; CIPN; Cryotherapy; Compression therapy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: The preferred intervention can be selected during the ongoing enrollment as soon as the pre-specified selection criteria are met, and further enrollment will cease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cryotherapy (Active Comparator): Men or women over the age of 18 with a history of stage I-III breast cancer and is scheduled to receive adjuvant or neoadjuvant paclitaxel or docetaxel for at least 12 weeks.
  Interventions: Device: Cryotherapy
- Compression Therapy (Active Comparator): Men or women over the age of 18 with a history of stage I-III breast cancer and is scheduled to receive adjuvant or neoadjuvant paclitaxel or docetaxel for at least 12 weeks.
  Interventions: Device: Compression Therapy
- Control arm (Loose glove/sock) (Placebo Comparator): Men or women over the age of 18 with a history of stage I-III breast cancer and is scheduled to receive adjuvant or neoadjuvant paclitaxel or docetaxel for at least 12 weeks.
  Interventions: Device: Loose glove/sock

INTERVENTIONS:
Device: Cryotherapy — Study subjects will wear NatraCure flexible socks on bilateral hands and feet. The sock will act as a mitten and covers the entire hand until past the wrist. There are 2 gel packs inserted into the sock, to provide cooling to the dorsal and frontal aspect of the hand. For the feet, the sock will cover the entire foot until above the ankle. Garments will be refrigerated for at least 3 hours at -25 to -30 Celsius prior to use. With each infusion, patients will wear the frozen garments on their hands and feet for a total of 90-120 minutes, beginning 15 minutes before the start of the infusion and until 15 minutes after the end of the infusion. Two sets of socks will be used during each session for 45-60 minutes each to maintain a consistently low temperatures of the extremities.
  Arms: Cryotherapy
Device: Compression Therapy — Study participants will wear Sigvaris Secure Arm Sleeves and Gloves on bilateral upper extremities. The sleeves and gloves provide 20-30mmHg of compression. Subjects will wear Sigvaris CompreFlex Lite compression garments on the lower extremities which includes a transition liner with a compressive foot, providing 20-30mmHg of compression on the lower leg and 15mmHg on the toes and feet. AccuTabs will be placed along the CompreFlex Lite to easily and accurately set the compression level at 20-30mmHg. With each chemotherapy infusion, patients will wear the sleeves/gloves and socks for a total of 90-120 minutes, beginning 15 minutes before the start of the infusion and until 15 minutes after the end of the infusion.
  Arms: Compression Therapy
Device: Loose glove/sock — Study participants will wear a non-compressive sleeve and loosely fitting glove on bilateral arms and hands. They will also wear a non-compressive Sigvaris Basic Liner with the CompreFlex Lite loosely applied over it. The investigators will verify that no compression is applied via using an interface pressure sensor (PicoPress). The maximum level of allowed pressure for garments will be 3mmHg. If the pressure reading is greater than 3mmHg, then a larger garment size will be used. Measurements with the pressure sensor will be repeated as needed to ensure a low pressure level of less than 3mmHg. With each chemotherapy infusion, patients will wear the gloves and socks for a total of 90-120 minutes, beginning 15 minutes before the start of the infusion and until 15 minutes after the end of the infusion.
  Arms: Control arm (Loose glove/sock)

SUMMARY:
The primary objective of this study is to select the best intervention from cold therapy, compression therapy and placebo at reducing neuropathic pain as measured by the change in the Neurotoxicity (NTX) component of the Functional Assessment of Cancer Therapy (FACT) - Taxane questionnaire, following 12 weeks of neoadjuvant/adjuvant chemotherapy with paclitaxel or docetaxel among breast cancer patients.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is a frequent side effect resulting from the administration of cytotoxic chemotherapeutic agents. The incidence of CIPN can vary on the type of agent used, the frequency with which it is given, and the cumulative dose. Unfortunately, for some patients, symptoms may persist even after discontinuation of the drug due to irreversible nerve damage. As of now, there are no established agents for CIPN prevention.

This is a randomized, placebo-controlled clinical selection trial of interventions for CIPN in patients treated with docetaxel every 3 weeks or paclitaxel on a weekly schedule. Patients will be randomly assigned to receive either frozen gloves and socks, compression gloves and socks, or "loose" gloves and socks (placebo arm) during chemotherapy infusion to study the best intervention at reducing neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years.
* History of stage I-III breast cancer
* Patient scheduled to be receiving adjuvant or neoadjuvant paclitaxel or docetaxel for at least 12 weeks
* Signed informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%,)

Exclusion Criteria:

* Prior treatment with taxane or platinum based chemotherapy
* Known history of neuropathy
* Raynaud's phenomenon
* Peripheral arterial ischemia
* Cold intolerance
* Current use of duloxetine which may mitigate chemotherapy-induced peripheral neuropathy (CIPN)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Accordino, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Accordino MK, Lee S, Leu CS, Levin B, Trivedi MS, Crew KD, Kalinsky K, Raghunathan R, Faheem K, Harden E, Taboada A, de Oliveira BD, Larson E, Franks L, Honan E, Law C, Hershman DL. Randomized adaptive selection trial of cryotherapy, compression therapy, and placebo to prevent taxane-induced peripheral neuropathy in patients with breast cancer. Breast Cancer Res Treat. 2024 Feb;204(1):49-59. doi: 10.1007/s10549-023-07172-y. Epub 2023 Dec 7. PMID 38060077

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Started | 20 | 22 | 21
Completed | 18 | 20 | 19
Not Completed | 2 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Death | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock) | Total
Number analyzed (Participants) | 20 | 22 | 21 | 63
Age, Continuous [Median (Full Range); unit: years] | 58.5 [36 to 82] | 53.5 [28 to 75] | 51.0 [34 to 78] | 53.5 [28 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 21 | 63
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 8 | 28
  Not Hispanic or Latino | 6 | 10 | 10 | 26
  Unknown or Not Reported | 3 | 3 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 4 | 15
  White | 5 | 6 | 7 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 7 | 5 | 21
Number docetaxel of treatments before baseline [Mean (Standard Deviation); unit: treatments] | 5.1 (1.3) | 5.5 (0.9) | 4.8 (1.7) | 5.1 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Successful Outcomes (<5-point Decrease in FACT-NTX From Baseline)
Description: The primary endpoint is the change in FACT NTX at 12 weeks from the start of chemotherapy. The change in FACT NTX will be dichotomized into a good outcome (change in FACT NTX less than 5 from baseline to week 12) versus a poor outcome (change in FACT NTX greater than or equal to 5 from baseline to week 12). The FACT-NTX subscale includes 11 items, each of which is divided into 5 scoring levels: 0, 1, 2, 3, 4, and a total score of 44. The scale is graded 0-4. A low score indicates a good effect. This change in FACT-NTX scale score indicates the proportion of patients with successful outcomes.
Time Frame: Baseline, 12 weeks
Measure: Number (95% Confidence Interval); unit: Proportion of Patients
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 20 | 22 | 21
Proportion of Patients | 0.45 [0.23 to 0.68] | 0.59 [0.36 to 0.79] | 0.52 [0.30 to 0.74]

2. Secondary Outcome: Change in NCI-CTCAE Grade for CIPN
Description: National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) is a subjective method to evaluate CIPN which is performed by a healthcare professional. The patient's peripheral sensory neuropathy, peripheral motor neuropathy, dysesthesia, paresthesia and neuralgia will be graded on a scale of 1 to 5 depending on severity with 1 indicating a better outcome.
Time Frame: Baseline, 12, and 24 weeks
Population: The numbers analyzed at the each of the respective timepoints are the number of participants from which the data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 18 | 21 | 19
Participants
  Week 12: number analyzed (Participants) | 16 | 21 | 18
  Week 12: Stage decreased | 1 | 0 | 1
  Week 12: Stage increased | 10 | 8 | 7
  Week 12: Stage stayed the same | 5 | 13 | 10
  Week 24: number analyzed (Participants) | 18 | 20 | 19
  Week 24: Stage decreased | 1 | 0 | 2
  Week 24: Stage increased | 11 | 8 | 7
  Week 24: Stage stayed the same | 6 | 12 | 10

3. Secondary Outcome: Change in Nail Toxicity
Description: The number of participants with a change in cutaneous toxicity and onycholysis will be assessed by a healthcare professional using the National Cancer Institute Common Toxicity Criteria (Version 2), specifically nail changes. Grade 1 includes discoloration, ridging (koilonychia), or pitting of the nails and Grade 2 is partial or complete loss of nail(s) or pain in the nail beds. A higher grade indicates more nail toxicity.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 14 | 15 | 16
Participants
  Week 12: Staged decreased | 0 | 0 | 1
  Week 12: Stage increased | 10 | 7 | 10
  Week 12: Stage stayed the same | 4 | 8 | 5
  Week 24: number analyzed (Participants) | 8 | 13 | 15
  Week 24: Staged decreased | 0 | 0 | 1
  Week 24: Stage increased | 7 | 7 | 11
  Week 24: Stage stayed the same | 1 | 6 | 3

4. Secondary Outcome: Comfort With Intervention Scale Score
Description: Comfort with the study intervention will be assessed on a 4-point scale, (0=dissatisfied; 1=not satisfied; 2=satisfied; 3=very satisfied) with 3 indicating a better outcome.
Time Frame: Up to 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 16 | 21 | 16
Participants
  Week 12: Dissatisfied | 4 | 2 | 0
  Week 12: Not Satisfied | 0 | 0 | 1
  Week 12: Satisfied | 9 | 13 | 12
  Week 12: Very Satisfied | 3 | 6 | 3
  Week 24: number analyzed (Participants) | 12 | 18 | 15
  Week 24: Dissatisfied | 3 | 1 | 0
  Week 24: Not Satisfied | 2 | 0 | 1
  Week 24: Satisfied | 5 | 10 | 11
  Week 24: Very Satisfied | 2 | 7 | 3

5. Secondary Outcome: Vibration Perception and Disappearance Threshold
Description: Study participants will be assessed for development of sensory neurological dysfunction. Vibration perception will be assessed using a tuning fork. Vibration threshold will be tested on the bilateral dorsum of the distal interphalangeal joint of the index finger and dorsum of the interphalangeal joint of the hallux. Subjects will be asked to indicate when the vibration stimulus is initially felt (perception threshold) and when the stimulus disappears (disappearance threshold.) The vibration perception threshold is the average of three paired measurements.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 20 | 22 | 21
Seconds
  Week 12: Hand Perception | 10.95 (7.34) | 7.70 (3.02) | 8.47 (4.72)
  Week 12: Foot Perception | 20.55 (13.13) | 17.16 (12.25) | 13.29 (6.29)
  Week 24: Hand Perception | 9.79 (6.28) | 7.82 (3.61) | 7.61 (2.30)
  Week 24: Foot Perception | 24.38 (18.54) | 20.84 (13.42) | 13.84 (5.56)
  Week 12: Hand Disapperance | 4.43 (3.87) | 3.09 (1.96) | 3.60 (4.02)
  Week 12: Foot Disappearance | 12.12 (9.53) | 11.33 (8.51) | 7.53 (5.54)
  Week 24: Hand Disappearance | 3.33 (3.39) | 3.04 (2.57) | 2.98 (2.23)
  Week 24: Foot Disappearance | 10.52 (6.15) | 12.90 (10.36) | 6.08 (3.91)

6. Secondary Outcome: Subjects Perceived Pain and Pressure Using Neuropen Test
Description: Evaluation of other sensory endpoints including touch, pressure and pain will be evaluated using a Neuropen. Touch and pressure sensation will be assessed using a 10-g monofilament on the subject's dominant foot. Pain and subjective sharpness sensation will be assessed using the Neuropen on the dominant foot. The spring mechanism is calibrated to exert a force of 40 grams to help identify subjects with loss of pain sensation. Ten points on the foot are tested. If the participant detects pain and pressure on less than 8 points, pain and pressure perception are considered diminished. Perception on 8 points of the foot or greater is considered a better outcome.
Time Frame: Up to 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 14 | 18 | 17
Participants
  Week 12: Touch and Pressure: number analyzed (Participants) | 14 | 18 | 13
  Week 12: Touch and Pressure: <8 points of the foot | 3 | 0 | 0
  Week 12: Touch and Pressure: >=8 points of the foot | 11 | 18 | 13
  Week 12: Pain: number analyzed (Participants) | 14 | 18 | 13
  Week 12: Pain: <8 points of the foot | 0 | 1 | 0
  Week 12: Pain: >=8 points of the foot | 14 | 17 | 13
  Week 24: Touch and Pressure: number analyzed (Participants) | 13 | 17 | 17
  Week 24: Touch and Pressure: <8 points of the foot | 3 | 0 | 0
  Week 24: Touch and Pressure: >=8 points of the foot | 10 | 17 | 17
  Week 24: Pain: number analyzed (Participants) | 13 | 17 | 17
  Week 24: Pain: <8 points of the foot | 1 | 0 | 0
  Week 24: Pain: >=8 points of the foot | 12 | 17 | 17

7. Secondary Outcome: Average Time to Complete 'Timed Get up and go' Test
Description: The 'timed get up and go' test is a rapid and widely used clinical performance-based measure of lower extremity function, mobility, and fall risk. Subjects are asked to stand up from a standard chair (seat height between 44 and 47 cm), walk a distance of 3 m (marked on the floor) at a comfortable pace, turn, walk back and sit down. Time will be measured in seconds. Shorter times indicate better performance.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 20 | 22 | 21
Seconds
  Week 12 | 15.48 (7.98) | 12.36 (3.75) | 15.18 (4.54)
  Week 24 | 17.45 (8.03) | 13.93 (3.04) | 14.84 (5.50)

8. Secondary Outcome: Tandem and Unipedal Stance Test
Description: Balance will be assessed using the tandem and unipedal stance test. In this assessment, the subject stands with one foot in front of the other (heel to toe) (30 seconds), then on one leg with: eyes open (60 seconds), eyes closed (30 seconds), and eyes open with head rotation (30 seconds) with arms held comfortably at the side. The test was accepted failure when the stance foot shifted in any way or the nonstance foot touched the ground. Tests are recorded as achieved (yes) or not achieved (no).
Time Frame: Up to 24 weeks
Population: The numbers analyzed at the each of the respective timepoints and assessments are the number of participants from which the data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 13 | 19 | 17
Participants
  Week 12: One leg, eyes open: number analyzed (Participants) | 13 | 19 | 15
  Week 12: One leg, eyes open: No | 6 | 12 | 11
  Week 12: One leg, eyes open: Yes | 7 | 7 | 4
  Week 12: One leg, eyes closed: number analyzed (Participants) | 13 | 19 | 15
  Week 12: One leg, eyes closed: No | 13 | 17 | 15
  Week 12: One leg, eyes closed: Yes | 0 | 2 | 0
  Week 12: One leg, eyes open, rotated: number analyzed (Participants) | 12 | 19 | 15
  Week 12: One leg, eyes open, rotated: No | 11 | 15 | 14
  Week 12: One leg, eyes open, rotated: Yes | 1 | 4 | 1
  Week 24: One leg, eyes open: number analyzed (Participants) | 13 | 16 | 17
  Week 24: One leg, eyes open: No | 10 | 11 | 11
  Week 24: One leg, eyes open: Yes | 3 | 5 | 6
  Week 24: One leg, eyes closed: number analyzed (Participants) | 13 | 16 | 17
  Week 24: One leg, eyes closed: No | 13 | 16 | 14
  Week 24: One leg, eyes closed: Yes | 0 | 0 | 3
  Week 24: One leg, eyes open, rotated: number analyzed (Participants) | 13 | 16 | 17
  Week 24: One leg, eyes open, rotated: No | 12 | 14 | 14
  Week 24: One leg, eyes open, rotated: Yes | 1 | 2 | 3

9. Secondary Outcome: Adherence to Study Intervention
Description: The number of participants who adhered to the intervention. Adherence is defined as wearing the assigned gloves and socks for greater than or equal to 80% of infusions.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
Number analyzed (Participants) | 20 | 22 | 21
Participants
  80% or Above | 7 | 16 | 16
  Below 80% | 13 | 6 | 5

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Cryotherapy | Compression Therapy | Control Arm (Loose Glove/Sock)
All-Cause Mortality (participants affected / at risk) | 0/20 | 2/22 | 1/21
Serious Adverse Events (participants affected / at risk) | 3/20 | 3/22 | 1/21
Other Adverse Events (participants affected / at risk) | 16/20 | 20/22 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy (N=20) | Compression Therapy (N=22) | Control Arm (Loose Glove/Sock) (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1) | 0 | 0
Confusion (Psychiatric disorders) | 1 (1) | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Urinary tract infection (Infections and infestations) | 0 | 1 (1) | 0
Fever (General disorders) | 0 | 1 (1) | 0
Non-cardiac chest pain (General disorders) | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryotherapy (N=20) | Compression Therapy (N=22) | Control Arm (Loose Glove/Sock) (N=21)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 9 (11) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 6 (6) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 8 (12) | 12 (12) | 6 (8)
Dysgeusia (Nervous system disorders) | 3 (4) | 8 (8) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Edema limbs (General disorders) | 4 (4) | 1 (1) | 3 (3)
Fatigue (General disorders) | 6 (7) | 13 (16) | 10 (10)
Administration site conditions (General disorders) | 3 (4) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 5 (5) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 7 (7)
Nail discoloration (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) | 10 (10)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 10 (11) | 12 (12) | 10 (11)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (5) | 3 (3) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5) | 4 (5)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT03873272/Prot_SAP_000.pdf